CLINICAL TRIAL: NCT01414322
Title: Documentation of Continuous Wheeze and Cough Dynamics in Pediatric ER SOB Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: KarmelSonix Ltd. (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Noam Gavriely, MD PhD, KarmelSonix Ltd.
Other Study IDs: KSI-IL-HHZ-ER-01
Record Dates: First submitted 2011-08-02; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Asthma; Bronchiolitis
MeSH Terms: conditions — Asthma; Bronchiolitis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Patients ages 0 - 3
- Group 2: Patients ages 3 - 7
- Group 3: Patients ages 7 - 15

SUMMARY:
Phenotype characterization of shortness of breath of pediatric emergency room patients by objective wheeze and cough monitoring improves diagnostic and severity assessment accuracy and correlates with overall patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patient is admitted to the ER with shortness of breath
* patient management is according to standardized protocols used in Hadassah Mt. Scopus pediatric emergency department including:

  * asthma management protocol
  * bronchiolitis management protocol
* ages 0 - 15
* patient's parent/guardian is able to comprehend and give informed consent for participating in the study

Exclusion Criteria:

* patient has received any dose of inhaled bronchodilators in the hour prior to enrollment
* patient has received oral or IV steroids in a time window of 30 minutes to 5 hours prior to enrollment
* ventilated patients, while ventilated
* chest skin lesions
* cystic fibrosis
* hemodynamic instability
* patient's parent/guardian objects to the study protocol
* concurrent participation in any other clinical study
* physician objection

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric emergency room patients ages 0 - 15 with shortness of breath upon arrival at the hospital
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-03 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
increase or decrease of WheezeRate (the proportion of wheezing in the respiratory cycle) | Duration (from beginning to end) of emergency department stay. On average, 3 hours.
  Characterize the dynamic pattern of wheeze rate (increase or decrease by 50% or unchanged) within 30 minutes of onset of therapy, and to correlate pattern to clinical diagnoses, severity assessment (accessory muscle use, oxygen saturation, inspiratory/expiratory ratio, severity of wheezing), and outcome (admission versus discharge).

SECONDARY OUTCOMES:
cough count (increase or decrease by more then 1 cough event or unchanged) in response to treatment | Duration (from beginning to end) of emergency department stay. On average, 3 hours.
  cough count (increase or decrease by more then 1 cough event or unchanged) in response to treatment and to correlate pattern to clinical diagnoses, severity assessment (accessory muscle use, oxygen saturation, inspiratory/expiratory ratio, severity of wheezing), and outcome (admission versus discharge).

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Kerem, Prof., Principal Investigator — Hadassah Medical Center Mt. Scopus, Jerusalem, Israel
Locations (1):
- Hadassah Medical Center Mt. Scopus, Jerusalem, Israel